CLINICAL TRIAL: NCT01482351
Title: Mild Cognitive Impairment and Obstructive Sleep Apnea
Acronym: MEMORIES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: George Mason University (Other)
Collaborators: National Institute on Aging (NIA) (NIH); University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Kathy C. Richards, University Professor, George Mason University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 7584; R01AG034682-01A2 (NIH)
Record Dates: First submitted 2011-11-28; First posted 2011-11-30 (Estimated); Results first posted 2019-01-29 (Actual); Last update posted 2019-03-06 (Actual); Status verified 2019-02

CONDITIONS: Obstructive Sleep Apnea; Mild Cognitive Impairment
Keywords: apnea; cognition; memory; function; amnestic mild cognitive impairment; older adults; Alzheimer's Disease
MeSH Terms: conditions — Sleep Apnea, Obstructive; Cognitive Dysfunction; Apnea; Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: Memories 1 was originally designed as a 6-month double-blind randomized controlled pilot trial of active versus placebo CPAP followed by a 6-month open label trial. However, after 1 year of recruitment of 371 individuals, no one consented to be randomized. Both older adults with MCI and their physicians perceived the placebo arm as an unnecessary risk. Although CPAP eliminates OSA, it must be consistently used for at least 4 hours per night for a therapeutic response, and only 30-60% of individuals prescribed CPAP adhere to it. The investigators, the study Data Safety Monitoring Board, and the NIH approved a change to a quasi-experimental study with 2 comparison groups: 1) an MCI, OSA, and CPAP adherent group (MCI+CPAP, ≥4 hr mean CPAP use per night for 1 year); and (2) an MCI, OSA, CPAP non-adherent group (MCI-CPAP, <4 hr mean CPAP use per night for 1 year). The final sample at 1 year consisted of 54 older adults with MCI: (1) MCI+CPAP, n = 29; and (2) MCI-CPAP, n = 25.
Who Masked: Outcomes Assessor
Masking Description: Persons collecting and analyzing neurocognitive data were blinded to participants' CPAP adherence.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MCI/OSA/CPAP Adherent (Experimental): Device: Continuous Positive Airway Pressure (CPAP). This arm included those diagnosed with mild cognitive impairment (MCI) and obstructive sleep apnea (OSA). The diagnostic criteria for OSA was defined as an Apnea Hypopnea Index (AHI) score of greater than or equal to 10. CPAP was prescribed for nightly use. Mean CPAP use in this arm was equal to or greater than 4 hours per night over one year. CPAP adherence Intervention was provided by research staff.
  Interventions: Behavioral: CPAP adherence intervention
- MCI/OSA/CPAP Non-adherent (Experimental): Device: Continuous Positive Airway Pressure (CPAP). This arm included those diagnosed with mild cognitive impairment (MCI) and obstructive sleep apnea (OSA). The diagnostic criteria for OSA was defined as an Apnea Hypopnea Index (AHI) score of greater than or equal to 10. CPAP was prescribed for nightly use. Mean CPAP use in this arm was less than 4 hours per night or CPAP use was withdrew for any reason over one year. Attention control intervention was provided by staff.
  Interventions: Behavioral: Attention control intervention

INTERVENTIONS:
Behavioral: CPAP adherence intervention — Critical factors were (1) OSA education, treatment expectations, and ways to minimize barriers and facilitate CPAP use; (2) promotion of a positive initial CPAP experience; (3) motivational interviewing to reinforce participants' health-related goals and CPAP self-efficacy; (4) anticipatory guidance and follow-up of common CPAP problems; and (5) social support by a study partner. Trained project staff provided the intervention by phone and face to face for a total of 12-14 hours over the 1 year project.
  Arms: MCI/OSA/CPAP Adherent
Behavioral: Attention control intervention — This intervention, provided by phone and face to face by project staff, provided equal time and attention. Critical factors were (1) education about OSA and risks, (2) education about memory, and other health topics of interest to the participants; (3) motivational interviewing to reinforce participants' health-related goals; (4) building rapport, and (5) social support by a study partner.
  Arms: MCI/OSA/CPAP Non-adherent

SUMMARY:
Obstructive sleep apnea (OSA) has been linked to increased risk for Alzheimer's disease (AD), but little prospective evidence exists on the effects of OSA treatment in preclinical AD. The objective was to determine if CPAP treatment adherence, controlling for baseline differences, predicts cognitive and everyday function after 1 year in older adults with MCI and to determine effect sizes for a larger trial. The aim of the Mild Cognitive Impairment and Obstructive Sleep Apnea (Memories 1) trial was to determine whether CPAP treatment adherence, controlling for any baseline differences in OSA severity, ApoE4, and other previously identified demographic and patient factors, might predict cognitive and everyday function after 1 year in older adults with amnestic MCI.

DETAILED DESCRIPTION:
In this prospective open label clinical trial, primary inclusions were age 55-89 years and apnea-hypopnea index ≥ 10. Groups were: (1) MCI, OSA, and CPAP adherent (MCI+CPAP); (2) MCI, OSA, CPAP nonadherent(MCI-CPAP). There were 68 MCI+OSA participants at baseline, and 14 (21%) dropped out during the 1 year follow-up. At 1 year, n=54, with MCI+CPAP group n=29, and MCI-CPAP group n=25. Statistically significant improvements in psychomotor/cognitive processing speed in the MCI+CPAP group versus the MCI-CPAP group were observed at 1 year after adjustment for age, race, and marital status. There were small to moderate effect sizes (ES) for memory, attention, daytime sleepiness, and everyday function, favoring the MCI+CPAP group versus the MCI-CPAP group.

ELIGIBILITY:
Inclusion criteria

Participants are included in the study if all of the following criteria are met:

(1) Are able to provide written informed consent by self or legally authorized representative. MacArthur Competency Assessment Tool for Clinical Research (MacCAT-CR) will be used to assess decision making capacity; (2) OSA defined as an apnea-hypopnea index (AHI) ≥10, using either a clinical split- or whole-night polysomnography. We chose an AHI cut-off of ≥10 as opposed to ≥15, the conventional cut-off for moderate OSA because split-night studies underestimate the AHI; (3) education-adjusted scores of 28-35 on the modified Telephone Interview for Cognitive Status; (4) 0-0.5 on the Clinical Dementia Rating (CDR); (5) 24-30 on the Mini-Mental State Examination (MMSE); (6) memory impairment approximately 1.0-1.5 standard deviations below normal (adjusted for age and education), determined by scores on the Logical Memory II test; (7) performance approximately 1.0-1.5 standard deviations below normal (adjusted for age and education) in no more than one cognitive domain in addition to memory; (8) medications stable for at least 4 weeks; washout from psychoactive medications (e.g., excluded anti-depressants, neuroleptics, chronic anxiolytics, and sedative hypnotics) for 4 weeks; (9) score of ≤28 on the 21-item Beck Depression Inventory II; (10) a study partner who spends at least 10 hours per week in phone or in-person contact with participant; (11) visual and auditory acuity for testing; (12) 6 or more grades of education completed, or a history to exclude intellectual disability; and (13) English fluency.

Exclusion criteria

Patients are excluded from participating in this study if 1 or more of the following criteria are met:

(1) significant neurologic disease other than MCI; (2) MRI exclusions, e.g. metal; (3) psychiatric disorders, including uncontrolled major depression, bipolar disorder, or schizophrenia; (4) history of alcohol dependence within 6 months; (5) current significant unstable medical condition; (6) participation in studies involving neuropsychological testing; (7) currently receiving CPAP; (8) requiring oxygen during CPAP; (9) dementia indicated by impairment in 3-5 age and education adjusted cognitive domains.

Ages: 55 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2012-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathy Richards, PhD, RN, Principal Investigator — George Mason University
Locations (3):
- United States (3):
  - Abington Memorial Hospital, Abington, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - George Mason University, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Data have been prepared for sharing with other investigators. Data can be accessed at http://dx.doi.org/10.15139/S3/12081 after publication of the main study findings.
Time Frame: Data will be made available 6 months after publication of the main study findings and will be available in perpetuity.
Access Criteria: Individual participant data (IPD) will be publicly available via the following url
URL: http://dx.doi.org/10.15139/S3/12081

REFERENCES:
- [Background] Terpening Z, Lewis SJ, Yee BJ, Grunstein RR, Hickie IB, Naismith SL. Association between Sleep-Disordered Breathing and Neuropsychological Performance in Older Adults with Mild Cognitive Impairment. J Alzheimers Dis. 2015;46(1):157-65. doi: 10.3233/JAD-141860. PMID 25720400
- [Background] Osorio RS, Gumb T, Pirraglia E, Varga AW, Lu SE, Lim J, Wohlleber ME, Ducca EL, Koushyk V, Glodzik L, Mosconi L, Ayappa I, Rapoport DM, de Leon MJ; Alzheimer's Disease Neuroimaging Initiative. Sleep-disordered breathing advances cognitive decline in the elderly. Neurology. 2015 May 12;84(19):1964-71. doi: 10.1212/WNL.0000000000001566. Epub 2015 Apr 15. PMID 25878183
- [Background] Guarnieri B, Adorni F, Musicco M, Appollonio I, Bonanni E, Caffarra P, Caltagirone C, Cerroni G, Concari L, Cosentino FI, Ferrara S, Fermi S, Ferri R, Gelosa G, Lombardi G, Mazzei D, Mearelli S, Morrone E, Murri L, Nobili FM, Passero S, Perri R, Rocchi R, Sucapane P, Tognoni G, Zabberoni S, Sorbi S. Prevalence of sleep disturbances in mild cognitive impairment and dementing disorders: a multicenter Italian clinical cross-sectional study on 431 patients. Dement Geriatr Cogn Disord. 2012;33(1):50-8. doi: 10.1159/000335363. Epub 2012 Mar 8. PMID 22415141
- [Background] Dzierzewski JM, Wallace DM, Wohlgemuth WK. Adherence to Continuous Positive Airway Pressure in Existing Users: Self-Efficacy Enhances the Association between Continuous Positive Airway Pressure and Adherence. J Clin Sleep Med. 2016 Feb;12(2):169-76. doi: 10.5664/jcsm.5478. PMID 26350607
- [Background] Sawyer AM, Gooneratne NS, Marcus CL, Ofer D, Richards KC, Weaver TE. A systematic review of CPAP adherence across age groups: clinical and empiric insights for developing CPAP adherence interventions. Sleep Med Rev. 2011 Dec;15(6):343-56. doi: 10.1016/j.smrv.2011.01.003. Epub 2011 Jun 8. PMID 21652236
- [Background] Khawaja IS, Olson EJ, van der Walt C, Bukartyk J, Somers V, Dierkhising R, Morgenthaler TI. Diagnostic accuracy of split-night polysomnograms. J Clin Sleep Med. 2010 Aug 15;6(4):357-62. PMID 20726284
- [Background] Petersen RC, Smith GE, Waring SC, Ivnik RJ, Tangalos EG, Kokmen E. Mild cognitive impairment: clinical characterization and outcome. Arch Neurol. 1999 Mar;56(3):303-8. doi: 10.1001/archneur.56.3.303. PMID 10190820
- [Background] Bennett DA, Wilson RS, Schneider JA, Evans DA, Beckett LA, Aggarwal NT, Barnes LL, Fox JH, Bach J. Natural history of mild cognitive impairment in older persons. Neurology. 2002 Jul 23;59(2):198-205. doi: 10.1212/wnl.59.2.198. PMID 12136057
- [Background] Rosness TA, Haugen PK, Engedal K. The clinical dementia rating scale could be helpful in differentiating frontotemporal dementia from Alzheimer's disease. Int J Geriatr Psychiatry. 2011 Aug;26(8):879-80. doi: 10.1002/gps.2555. No abstract available. PMID 21744389
- [Background] Crum RM, Anthony JC, Bassett SS, Folstein MF. Population-based norms for the Mini-Mental State Examination by age and educational level. JAMA. 1993 May 12;269(18):2386-91. PMID 8479064
- [Background] Morris J, Swier-Vosnos A, Woodworth C, Umfleet LG, Czipri S, Kopald B. Development of alternate paragraphs for the Logical Memory subtest of the Wechsler Memory Scale-IV. Appl Neuropsychol Adult. 2014;21(2):143-7. doi: 10.1080/09084282.2013.780172. Epub 2013 Sep 11. PMID 24826508
- [Background] Wang YP, Gorenstein C. Psychometric properties of the Beck Depression Inventory-II: a comprehensive review. Braz J Psychiatry. 2013 Oct-Dec;35(4):416-31. doi: 10.1590/1516-4446-2012-1048. Epub 2013 Dec 23. PMID 24402217
- [Background] Kapur VK, Auckley DH, Chowdhuri S, Kuhlmann DC, Mehra R, Ramar K, Harrod CG. Clinical Practice Guideline for Diagnostic Testing for Adult Obstructive Sleep Apnea: An American Academy of Sleep Medicine Clinical Practice Guideline. J Clin Sleep Med. 2017 Mar 15;13(3):479-504. doi: 10.5664/jcsm.6506. PMID 28162150
- [Background] Basner M, Dinges DF. Maximizing sensitivity of the psychomotor vigilance test (PVT) to sleep loss. Sleep. 2011 May 1;34(5):581-91. doi: 10.1093/sleep/34.5.581. PMID 21532951
- [Background] Tomaszewski Farias S, Mungas D, Harvey DJ, Simmons A, Reed BR, Decarli C. The measurement of everyday cognition: development and validation of a short form of the Everyday Cognition scales. Alzheimers Dement. 2011 Nov;7(6):593-601. doi: 10.1016/j.jalz.2011.02.007. PMID 22055976
- [Background] Billings ME, Rosen CL, Auckley D, Benca R, Foldvary-Schaefer N, Iber C, Zee PC, Redline S, Kapur VK. Psychometric performance and responsiveness of the functional outcomes of sleep questionnaire and sleep apnea quality of life instrument in a randomized trial: the HomePAP study. Sleep. 2014 Dec 1;37(12):2017-24. doi: 10.5665/sleep.4262. PMID 25325491
- [Background] Schwartz SW, Sebastiao Y, Rosas J, Iannacone MR, Foulis PR, Anderson WM. Racial disparity in adherence to positive airway pressure among US veterans. Sleep Breath. 2016 Sep;20(3):947-55. doi: 10.1007/s11325-016-1316-1. Epub 2016 Jan 25. PMID 26810493
- [Background] Hakansson K, Rovio S, Helkala EL, Vilska AR, Winblad B, Soininen H, Nissinen A, Mohammed AH, Kivipelto M. Association between mid-life marital status and cognitive function in later life: population based cohort study. BMJ. 2009 Jul 2;339:b2462. doi: 10.1136/bmj.b2462. PMID 19574312
- [Background] Weaver TE, Grunstein RR. Adherence to continuous positive airway pressure therapy: the challenge to effective treatment. Proc Am Thorac Soc. 2008 Feb 15;5(2):173-8. doi: 10.1513/pats.200708-119MG. PMID 18250209
- [Background] Zimmerman ME, Arnedt JT, Stanchina M, Millman RP, Aloia MS. Normalization of memory performance and positive airway pressure adherence in memory-impaired patients with obstructive sleep apnea. Chest. 2006 Dec;130(6):1772-8. doi: 10.1378/chest.130.6.1772. PMID 17166995
- [Derived] Richards KC, Gooneratne N, Dicicco B, Hanlon A, Moelter S, Onen F, Wang Y, Sawyer A, Weaver T, Lozano A, Carter P, Johnson J. CPAP Adherence May Slow 1-Year Cognitive Decline in Older Adults with Mild Cognitive Impairment and Apnea. J Am Geriatr Soc. 2019 Mar;67(3):558-564. doi: 10.1111/jgs.15758. Epub 2019 Feb 6. PMID 30724333

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From 9/2012 to 12/2014, study investigators identified potential participants from clinical practices, advertisements in newspapers, clinical trials registries, senior centers, advertisements in public transportation centers, the Alzheimer's Association, and support groups.
Groups:
- Experimental: MCI/OSA/CPAP Adherent and Non-adherent: All participants were diagnosed with MCI and OSA. The diagnostic criteria for OSA was defined as an AHI score greater than or equal to 10. CPAP was prescribed for nightly use. At baseline there were 68 participants had OSA (AHI ≥10). 14 persons withdrew prior to 6 month testing. There were 54 active MCI participants with OSA at 6 months and 12 month: 29 were CPAP adherent and 25 were CPAP non-adherent.
Period: Overall Study
Arm/Group | Experimental: MCI/OSA/CPAP Adherent and Non-adherent
Started | 68
6 Months | 54 (14 dropped out)
12 Months | 54
Completed | 54
Not Completed | 14

BASELINE CHARACTERISTICS:
Population: Demographics, clinical characteristics and sleep data were described for the MCI/OSA/CPAP Adherent and MCI/OSA/CPAP non-adherent groups defined at 6 months using data from baseline (entry into study).
Groups:
- MCI/OSA/CPAP Adherent: Device: Continuous Positive Airway Pressure [CPAP]. Included those diagnosed with mild cognitive impairment (MCI) and obstructive sleep apnea (OSA). The diagnostic criteria for OSA was defined as an Apnea Hypopnea Index (AHI) score of greater than or equal to 10. CPAP was prescribed for nightly use. Mean CPAP use equal to or greater than 4 hours per night over one year.
  Continuous Positive Airway Pressure [CPAP]: Study participants with sleep apnea will choose to use or not use a continuous positive airway pressure (CPAP) machine to treat their apnea after a consultation with their doctor. Dosage of CPAP will be individually determined using standardized methods in an overnight CPAP titration polysomnography.
- MCI/OSA/CPAP Non-adherent: Device: Continuous Positive Airway Pressure [CPAP]. Included those diagnosed with mild cognitive impairment (MCI) and obstructive sleep apnea (OSA). The diagnostic criteria for OSA was defined as an Apnea Hypopnea Index (AHI) score of greater than or equal to 10. CPAP was prescribed for nightly use. Mean CPAP use less than 4 hours per night over one year.
  Continuous Positive Airway Pressure [CPAP]: Study participants with sleep apnea will choose to use or not use a continuous positive airway pressure (CPAP) machine to treat their apnea after a consultation with their doctor. Dosage of CPAP will be individually determined using standardized methods in an overnight CPAP titration polysomnography.
- Total: Total of all reporting groups
Arm/Group | MCI/OSA/CPAP Adherent | MCI/OSA/CPAP Non-adherent | Total
Number analyzed (Participants) | 29 | 25 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.4 (7.2) | 73.2 (8.6) | 70.1 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 15 | 24
  Male | 20 | 10 | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 13 | 17
  White | 24 | 11 | 35
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 29 | 25 | 54
Education [Number; unit: participants] — Participants who have more than a high school education.
  participants | 26 | 21 | 47
Married/Cohabitate [Number; unit: participants] — Participants who are married or cohabitate.
  participants | 23 | 8 | 31
BMI [Mean (Standard Deviation); unit: kg/m^2] — Body mass index (BMI) is defined as the body mass divided by the square of the body height, and is expressed in units of kg/m2.
  kg/m^2 | 30.3 (6.7) | 29.5 (6.5) | 29.9 (6.6)
Income - <$20,000 [Count of Participants; unit: Participants] — Population: Only 45 of the 54 participants provided income data.
  Participants
    number analyzed (Participants) | 24 | 21 | 45
    (all) | 3 | 9 | 12
Income - $20,000 - $39,999 [Count of Participants; unit: Participants] — Population: Only 45 of the 54 participants provided income data.
  Participants
    number analyzed (Participants) | 24 | 21 | 45
    (all) | 2 | 2 | 4
Income - $40,000 - $69,999 [Count of Participants; unit: Participants] — Population: Only 45 of the 54 participants provided income data.
  Participants
    number analyzed (Participants) | 24 | 21 | 45
    (all) | 3 | 4 | 7
Income - $70,000 - $99,999 [Count of Participants; unit: Participants] — Population: Only 45 of the 54 participants provided income data.
  Participants
    number analyzed (Participants) | 24 | 21 | 45
    (all) | 4 | 2 | 6
Income - >$100,000 [Count of Participants; unit: Participants] — Population: Only 45 of the 54 participants provided income data.
  Participants
    number analyzed (Participants) | 24 | 21 | 45
    (all) | 12 | 4 | 16
Study Partner-Spouse/cohabitate [Count of Participants; unit: Participants] | 26 | 9 | 35
Study Partner-Adult child [Count of Participants; unit: Participants] | 1 | 6 | 7
Study Partner-Other [Count of Participants; unit: Participants] | 2 | 10 | 12
Reported/known conditions-Diabetes [Count of Participants; unit: Participants] | 7 | 8 | 15
Reported/known conditions-Cardiovascular Disease [Count of Participants; unit: Participants] | 11 | 14 | 25
Reported/known conditions-Hypertension [Count of Participants; unit: Participants] | 15 | 14 | 29
Apolipoprotein E (ApoE)-E2/E2 [Count of Participants; unit: Participants] — The Apolipoprotein E (ApoE) gene has three major forms: ApoE2, ApoE3 and ApoE4. The ApoE4 allele has been linked to higher incidence of development of Alzheimer's Disease (AD) as well as Obstructive Sleep Apnea (OSA). Population: Only 52 of the 54 participants provided data.
  Participants
    number analyzed (Participants) | 27 | 25 | 52
    (all) | 0 | 1 | 1
ApoE-E2/E3 [Count of Participants; unit: Participants] — The ApoE gene has three major forms: ApoE2, ApoE3 and ApoE4. The ApoE4 allele has been linked to higher incidence of development of AD as well as OSA. Population: Only 52 of the 54 participants provided data.
  Participants
    number analyzed (Participants) | 27 | 25 | 52
    (all) | 1 | 0 | 1
ApoE-E2/E4 [Count of Participants; unit: Participants] — The ApoE gene has three major forms: ApoE2, ApoE3 and ApoE4. The ApoE4 allele has been linked to higher incidence of development of AD as well as OSA. Population: Only 52 of the 54 participants provided data.
  Participants
    number analyzed (Participants) | 27 | 25 | 52
    (all) | 1 | 0 | 1
ApoE-E3/E3 [Count of Participants; unit: Participants] — The ApoE gene has three major forms: ApoE2, ApoE3 and ApoE4. The ApoE4 allele has been linked to higher incidence of development of AD as well as OSA. Population: Only 52 of the 54 participants provided data.
  Participants
    number analyzed (Participants) | 27 | 25 | 52
    (all) | 16 | 18 | 34
ApoE-E3/E4 [Count of Participants; unit: Participants] — The ApoE gene has three major forms: ApoE2, ApoE3 and ApoE4. The ApoE4 allele has been linked to higher incidence of development of AD as well as OSA. Population: Only 52 of the 54 participants provided data.
  Participants
    number analyzed (Participants) | 27 | 25 | 52
    (all) | 9 | 4 | 13
ApoE-E4/E4 [Count of Participants; unit: Participants] — The ApoE gene has three major forms: ApoE2, ApoE3 and ApoE4. The ApoE4 allele has been linked to higher incidence of development of AD as well as OSA. Population: Only 52 of the 54 participants provided data.
  Participants
    number analyzed (Participants) | 27 | 25 | 52
    (all) | 0 | 2 | 2
Medications-Cholinesterase inhibitors [Count of Participants; unit: Participants] — An acetylcholinesterase inhibitor or anti-cholinesterase is a chemical or a drug that inhibits the acetylcholinesterase enzyme from breaking down acetylcholine, thereby increasing both the level and duration of action of the neurotransmitter acetylcholine.
  Participants | 1 | 2 | 3
Medications-NMDA Receptor Antagonist [Count of Participants; unit: Participants] — N-Methyl-D-aspartate (NMDA) receptor antagonists are a class of anesthetics that work to antagonize, or inhibit the action of, the NMDA receptor.
  Participants | 0 | 0 | 0
Medications-Opioid Analgesics [Count of Participants; unit: Participants] | 0 | 3 | 3
Medications-Antidepressants [Count of Participants; unit: Participants] | 6 | 1 | 7
Medications-Sedatives/anxiolytics [Count of Participants; unit: Participants] | 5 | 5 | 10
Medications-Antihypertensives [Count of Participants; unit: Participants] | 19 | 21 | 40
Medications-Cholesterol medications [Count of Participants; unit: Participants] | 21 | 18 | 39
MMSE [Mean (Standard Deviation); unit: units on a scale] — Mini-Mental State Examination (MMSE), a 30-point questionnaire with possible total scores ranging from 0-30 (higher scores are better). Inclusion criteria included normal general cognition defined as MMSE greater than or equal to 24.
  units on a scale | 28.3 (1.4) | 28.0 (2.1) | 28.2 (1.7)
CDR [Mean (Standard Deviation); unit: units on a scale] — Clinical Dementia Rating (CDR), a 5-point scale used to characterize six domains of cognitive and functional performance applicable to Alzheimer disease and related dementias (lower scores are better). 0 = Normal, 0.5 = Very Mild Dementia,1 = Mild Dementia, 2 = Moderate Dementia, 3 = Severe Dementia.
  units on a scale | 0.5 (0.3) | 0.7 (0.7) | 0.6 (0.5)
ESS [Mean (Standard Deviation); unit: units on a scale] — Epworth Sleepiness Scale (ESS) is an 8-item measure used to assess daytime sleepiness. Scores range from 0 to 24. Lower scores are better - indicating sleepiness is affecting functioning less.
  units on a scale | 8.5 (3.5) | 9.3 (5.3) | 8.9 (4.4)
BDI-II [Mean (Standard Deviation); unit: units on a scale] — Beck Depression Inventory Second Edition (BDI)-II is a 21-item instrument intended to assess the existence and intensity of symptoms of depression. Cut score guidelines for the BDI-II are given with the recommendation that thresholds be adjusted based on the characteristics of the sample, and the purpose for use of the BDI-II. Total score of 0-13 is considered minimal range, 14-19 is mild, 20-28 is moderate, and 29-63 is severe.
  units on a scale | 7.7 (4.6) | 6.4 (6.6) | 7.1 (5.6)
ARES - Total sleep time [Mean (Standard Deviation); unit: minutes] — Total sleep time assessed with the Apnea Risk Evaluation System (ARES), which is used to screen for sleep apnea.
  minutes | 441.0 (107.0) | 334.2 (35.6) | 374.3 (84.0)
ARES - Apnea-Hypopnea Index [Mean (Standard Deviation); unit: events/hour] — Apnea-Hypopnea Index (AHI) is assessed with the Apnea Risk Evaluation System (ARES), which is used to screen for sleep apnea. AHI is calculated by dividing the number of apnea events by the number of hours of sleep. AHI values for adults are categorized as: Normal: AHI<5; Mild sleep apnea: 5</=AHI<15; Moderate sleep apnea: 15</=AHI<30; Severe sleep apnea: AHI>/=30
  events/hour | 21.3 (7.8) | 14.6 (2.7) | 17.1 (5.8)
ARES - Lowest oxygen saturation [Mean (Standard Deviation); unit: percentage of blood oxygen saturation] — Lowest oxygen saturation assessed with the Apnea Risk Evaluation System (ARES), which is used to screen for sleep apnea. Normal blood oxygen levels in humans are considered 95-100 percent.
  percentage of blood oxygen saturation | 83.6 (4.3) | 82.9 (2.8) | 83.1 (3.1)
PSG - Total sleep time [Mean (Standard Deviation); unit: minutes] — Total sleep time assessed with polysomnography (PSG), also called a sleep study, which is used to diagnose sleep disorders.
  minutes | 283.2 (84.0) | 270.5 (95.9) | 279.0 (86.7)
PSG - Apnea-Hypopnea Index [Mean (Standard Deviation); unit: events/hour] — AHI assessed with polysomnography (PSG), also called a sleep study, which is used to diagnose sleep disorders. AHI is calculated by dividing the number of apnea events by the number of hours of sleep. AHI values for adults are categorized as: Normal: AHI<5; Mild sleep apnea: 5</=AHI<15; Moderate sleep apnea: 15</=AHI<30; Severe sleep apnea: AHI>/=30
  events/hour | 25.3 (11.5) | 31.1 (20.8) | 27.2 (15.0)
PSG - Lowest oxygen saturation [Mean (Standard Deviation); unit: percentage of blood oxygen saturation] — Lowest oxygen saturation assessed with polysomnography (PSG), also called a sleep study, which is used to diagnose sleep disorders. Normal blood oxygen levels in humans are considered 95-100 percent.
  percentage of blood oxygen saturation | 82.3 (6.9) | 81.8 (5.0) | 82.2 (6.3)
Split-night PSG - Total sleep time [Mean (Standard Deviation); unit: minutes] — Total sleep time assessed with split-night polysomnography (PSG), a strategy that encompasses both diagnosis of OSA and initiation of positive pressure therapy in a single night.
  minutes | 218.2 (150.6) | 150.4 (77.4) | 166.1 (95.7)
Split-night PSG - Apnea-Hypopnea index [Mean (Standard Deviation); unit: events/hour] — AHI assessed with split-night polysomnography (PSG), a strategy that encompasses both diagnosis of OSA and initiation of positive pressure therapy in a single night. AHI is calculated by dividing the number of apnea events by the number of hours of sleep. AHI values for adults are categorized as: Normal: AHI<5; Mild sleep apnea: 5</=AHI<15; Moderate sleep apnea: 15</=AHI<30; Severe sleep apnea: AHI>/=30
  events/hour | 25.6 (9.2) | 14.6 (7.8) | 17.7 (9.4)
Split-night PSG - Lowest oxygen saturation [Mean (Standard Deviation); unit: percentage of blood oxygen saturation] — Lowest oxygen saturation assessed with split-night polysomnography (PSG), a strategy that encompasses both diagnosis of OSA and initiation of positive pressure therapy in a single night. Normal blood oxygen levels in humans are considered 95-100 percent.
  percentage of blood oxygen saturation | 86.0 (5.0) | 82.9 (6.3) | 83.8 (6.0)

OUTCOME MEASURES:

1. Primary Outcome: Hopkins Verbal Learning Test-Revised (HVLT-R)
Description: Memory (immediate and delayed recall) will be assessed using HVLT-R. HVLT-R has been used in elders with Alzheimer's Disease and takes 10 minutes to complete. Total score ranges from 0 to 60, a higher score indicates a better memory (better outcome).
Time Frame: Change from baseline at 6 months and 1 year
Population: 14 participants lost to follow-up prior to 6-months testing.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- MCI/OSA/CPAP Non-adherent: Device: Continuous Positive Airway Pressure [CPAP]. Included those diagnosed with mild cognitive impairment (MCI) and obstructive sleep apnea (OSA). The diagnostic criteria for OSA was defined as an Apnea Hypopnea Index (AHI) score of greater than or equal to 10. CPAP prescribed for nightly use. Mean CPAP use less than 4 hours per night over one year.
  Continuous Positive Airway Pressure [CPAP]: Study participants with sleep apnea will choose to use or not use a continuous positive airway pressure (CPAP) machine to treat their apnea after a consultation with their doctor. Dosage of CPAP will be individually determined using standardized methods in an overnight CPAP titration polysomnography.
Arm/Group | MCI/OSA/CPAP Adherent | MCI/OSA/CPAP Non-adherent
Number analyzed (Participants) | 29 | 25
score on a scale
  Baseline | 23.52 (5.56) | 20.04 (5.30)
  6-month | 23.68 (5.08) | 20.39 (5.48)
  1 year: number analyzed (Participants) | 29 | 22
  1 year | 23.59 (5.73) | 20.82 (5.69)

2. Primary Outcome: Digit Symbol Subtest (DS)
Description: The Digit Symbol subtest (DS) from the Wechsler Adult Intelligence Scale (WAIS-R) was used to measure psychomotor/cognitive processing speed. An age-adjusted total scaled score was used for analysis. The adjusted total score ranges from -5.7 to+27. A higher score indicates a better outcome.
Time Frame: Change from baseline at 6 months and 1 year
Population: 14 participants lost to follow-up prior to 6-months testing.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MCI/OSA/CPAP Adherent | MCI/OSA/CPAP Non-adherent
Number analyzed (Participants) | 29 | 25
score on a scale
  Baseline | 9.18 (2.59) | 8.06 (2.65)
  6-months | 9.90 (2.74) | 8.02 (2.36)
  1 year: number analyzed (Participants) | 29 | 22
  1 year | 10.21 (3.03) | 8.09 (2.78)

3. Primary Outcome: Mini Mental State Evaluation Exam (MMSE)
Description: Global cognitive function will be assessed using MMSE. It is a 30-item cognitive screen measuring orientation, registration, short-term memory, attention/concentration, language, and constructional capacity. Summary score will be used as a measure of global cognitive function. Total score ranges from 0 to 30, equal to and above 24 is normal (better outcome), less than 21 indicates increasing odds of dementia (worse outcome).
Time Frame: Change from baseline at 6 months and 1 year
Population: 14 participants lost to follow-up prior to 6-months testing.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MCI/OSA/CPAP Adherent | MCI/OSA/CPAP Non-adherent
Number analyzed (Participants) | 29 | 25
score on a scale
  Baseline | 28.34 (1.40) | 28.00 (2.10)
  6-month | 28.61 (1.62) | 27.48 (2.00)
  1-year: number analyzed (Participants) | 29 | 22
  1-year | 27.93 (2.05) | 26.43 (2.46)

4. Primary Outcome: Stroop Color and Word Test (SCW)
Description: Attention will be measured using SCW. We used the Golden and Freshwater's (2002) version. This version provides paper stimuli for each trial: in the first, columns of the words"red""blue" and "green" are printed in black ink (Word Reading; W); in the second, columns of the same words are printed in red, blue, or green ink (Color Naming; C); in the third, the words "red" "blue" and "green" are printed in a colored ink (red, blue or green) that does not match the word (Color-Word; CW). Participants read each page aloud as quickly as possible for 45 seconds and receive a score for each trial representing the number of items correctly read aloud. The Interference T-score is obtained by first calculating a deviation score by subtracting a predicted CW score from the obtained raw CW score (in 45s). The obtained deviation score is then converted to an Interference T-score. Lower T scores(T<40) in the Interference condition show reductions in inhibitory control.
Time Frame: Change from baseline at 6 months and 1 year
Population: 14 participants were lost to follow-up prior to 6-months testing.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MCI/OSA/CPAP Adherent | MCI/OSA/CPAP Non-adherent
Number analyzed (Participants) | 29 | 25
score on a scale
  Baseline | 47.36 (6.15) | 44.28 (8.19)
  6-month | 48.22 (8.20) | 45.36 (8.57)
  1-year: number analyzed (Participants) | 29 | 22
  1-year | 50.00 (7.40) | 45.14 (9.47)

5. Primary Outcome: The Psychomotor Vigilance Task (PVT)
Description: Attention/reaction time will assessed using the PVT. The participants sat in a closed and quiet examination room, without any auditory or visual disturbance. A 1-minute mock PVT demonstration was done prior to each test. The PVT visual display was held 14-22 inches from the subject's eyes. The participants were asked to either use the index finger or thumb of their dominant hand to respond to the PVT signals. The participants were instructed to maintain the fastest possible reaction times to a simple visual stimulus: a red light emitting diode displaying time in milliseconds in a window of the portable PVT device. We used number of lapses, defined as mean reaction time above 500 milliseconds (errors of omission) as the primary outcome. Lower score indicates better outcomes (Less lapses).
Time Frame: Change from baseline at 6 months and 1 year
Population: 14 participants were lost to follow-up prior to 6-months testing.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MCI/OSA/CPAP Adherent | MCI/OSA/CPAP Non-adherent
Number analyzed (Participants) | 29 | 25
score on a scale
  Baseline | 3.09 (1.53) | 6.46 (3.66)
  6-month | 2.58 (1.64) | 4.29 (2.71)
  1-year | 2.77 (1.91) | 4.76 (2.94)

6. Primary Outcome: Epworth Sleepiness Scale [ESS]
Description: Daytime sleepiness be assessed using ESS. The ESS asks the respondent to rate the likelihood of falling asleep in eight specific situations using a four-point Likert scale ranging from never dozing to high chance of dozing. The scale significantly correlates with the frequency of apneas and is a clinical and research standard for the assessment of daytime sleepiness. The total score ranges from 0 to 24, a higher score indicates higher chance of daytime sleepiness (worse outcome).
Time Frame: Change from baseline at 6 months and 1 year
Population: 14 participants were lost to follow-up prior to 6-months testing.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MCI/OSA/CPAP Adherent | MCI/OSA/CPAP Non-adherent
Number analyzed (Participants) | 29 | 25
score on a scale
  Baseline | 8.50 (3.52) | 9.32 (5.34)
  6-months | 6.54 (3.17) | 8.00 (5.53)
  1-year: number analyzed (Participants) | 29 | 22
  1-year | 6.34 (3.71) | 7.57 (4.37)

7. Secondary Outcome: Functional Outcomes Sleep Questionnaire (FOSQ)
Description: Everyday function will be assessed using FOSQ. It is a 30-item Likert-scale, self-report, disease-specific functional status measure written at the 4th grade level. The total score ranges from 0 to 120, a higher score indicates a better outcome.
Time Frame: Change from baseline at 6 months and 1 year
Population: 14 participants were lost to follow-up prior to 6-months testing.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MCI/OSA/CPAP Adherent | MCI/OSA/CPAP Non-adherent
Number analyzed (Participants) | 29 | 25
score on a scale
  Baseline | 17.31 (1.99) | 17.34 (2.66)
  6-month | 18.17 (1.48) | 18.13 (2.14)
  1-year: number analyzed (Participants) | 29 | 22
  1-year | 18.30 (1.82) | 18.63 (1.95)

8. Secondary Outcome: Everyday Function Outcome: Everyday Cognition (E-Cog)
Description: This informant-rated composes of multiple subscales, to evaluate cognitively based functional abilities in older adults. The factor structure of Everyday Cognition was assessed with confirmatory factor analysis, which supported a 7-factor model including 1 global factor and 6 domain-specific factors (Everyday Memory, Language, Visuospatial Abilities, Planning, Organization, and Divided Attention). The total mean score ranges from 0 to 57. A higher score indicates a worse outcome.
Time Frame: Change from baseline at 6 months and 1 year
Population: 14 participants were lost to follow up prior to 6 months testing.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MCI/OSA/CPAP Adherent | MCI/OSA/CPAP Non-adherent
Number analyzed (Participants) | 29 | 25
score on a scale
  Baseline | 1.46 (0.54) | 1.29 (0.41)
  6 months | 1.35 (0.36) | 1.43 (0.52)
  1-year | 1.35 (0.51) | 1.52 (0.70)

9. Secondary Outcome: Alzheimer's Disease Cooperative Study - Clinicians' Global Impression of Change Scale (ADCS-CGIC)
Description: Global change (progression) will be assessed using ADCS-CGIC at 1 year. It has 8 categories as markedly improved, moderately improved, minimally improved, not changed, minimally worse, moderately worse, markedly worse, missing response.
Time Frame: Change from baseline at 1 year
Population: Participants who completed the study and improved on ADCS-CGIC scores at 1year adjusted for age, race and marital status.
Measure: Number; unit: participants
Groups:
- MCI-OSA: Participants who completed the study and had Alzheimer's Disease Clinician's Scale (ADCS) data adjusted for age, race, and marital status.
Arm/Group | MCI-OSA
Number analyzed (Participants) | 41
participants
  ADCS-CGIC Improved | 34
  ADCS-CGIC Unimproved | 7

10. Secondary Outcome: Clinical Dementia Rating Scale (CDR)
Description: Cognitive ability will be assessed and staged using CDR. It contains 6 items (memory, orientation, judgement and problem solving, community affairs, home and hobbies, personal care), and each item ranges from 0 to 3. The total score ranges from 0 to 18, a higher score indicates a worse outcome. We observed the change of CDR score from baseline to 1-year follow up. Improved on CDR was defined as a lower CDR score compared to baseline. Reference group is unimproved, defined as worsened (higher) CDR or unchanged CDR compared to baseline.
Time Frame: Change from baseline at 1 year
Population: Study participants who completed the study and improved on CDR data adjusted for age, race and marital status.
Measure: Number; unit: participants
Groups:
- MCI-OSA: Participants who completed the study and had Clinical Dementia Rating data.
Arm/Group | MCI-OSA
Number analyzed (Participants) | 42
participants
  CDR Improved | 21
  CDR Unimproved | 21

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- MCI/OSA/CPAP Adherent: Device: CPAP. Included those diagnosed with MCI and OSA. The diagnostic criteria for OSA was defined as an AHI score of greater than or equal to 10. CPAP was prescribed for nightly use. Mean CPAP use equal to or greater than 4 hours per night over one year.
- MCI/OSA/CPAP Non-adherent: Device: CPAP. Included those diagnosed with MCI and OSA. The diagnostic criteria for OSA was defined as an AHI score of greater than or equal to 10. CPAP was prescribed for nightly use. Mean CPAP use less than 4 hours per night over one year.
Arm/Group | MCI/OSA/CPAP Adherent | MCI/OSA/CPAP Non-adherent
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/25
Serious Adverse Events (participants affected / at risk) | 5/29 | 0/25
Other Adverse Events (participants affected / at risk) | 0/29 | 0/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MCI/OSA/CPAP Adherent (N=29) | MCI/OSA/CPAP Non-adherent (N=25)
Heart irregularities (Cardiac disorders) | 2 (2) | 0 (0) — Heart irregularities during polysomnography
Hospital admission (General disorders) | 1 (1) | 0 (0) — Hospital admission due to fall
Bleeding (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Bleeding post testosterone implant
Surgery (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Herniated disc surgery

LIMITATIONS AND CAVEATS:
The study was not a randomized double-blind trial, and the sample is small. The groups may have been different on unidentified variables, and it is possible that these differences affected the study outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No